CLINICAL TRIAL: NCT04955067
Title: Deep Learning of Anterior Talofibular Ligament: Comparison of Different Models
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2020460
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Lateral Ligament, Ankle
Keywords: artificial intelligence; anterior talofibular ligament; sports Injury
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal control group-Grade 0: Arthroscopic examination of the ankle joint was normal, and the ligament was intact without injury or tear.
  Interventions: Diagnostic Test: Diagnositic test
- Ligament injury -Grade 1: Arthroscopic examination of the ankle joint showed ligament degeneration or injury, but no local or complete tear.
  Interventions: Diagnostic Test: Diagnositic test
- Ligament tear-Grade 2: Arthroscopy of the ankle joint revealed partial or complete loss of ligaments.
  Interventions: Diagnostic Test: Diagnositic test

INTERVENTIONS:
Diagnostic Test: Diagnositic test — The results of hip arthroscopy were taken as the gold standard, and MRI examination was taken as the research object

SUMMARY:
The purpose of this study is to study the injury of the anterior talofibular ligament by deep learning method and compare a variety of different deep learning models to establish a deep learning method that can accurately identify and grade the injury of anterior talofibular ligament, and obtain a model with better recognition and grading effect.

DETAILED DESCRIPTION:
1. Recognition and segmentation of anterior talofibular ligament based on DenseNet. Densenet was used to recognize the axial T2-fs image, and the image level was the most typical one. The labelimg program based on Python was used to locate the coordinates of the anterior talofibular ligament and then imported into Python for learning. All the data were divided into a training set (70%, and then 30% of the training set was selected as the verification set). The remaining 30% was used as the test set to evaluate the accuracy of model recognition. After identifying the anterior talofibular ligament, the local clipping and amplification are carried out to remove the redundant information. Finally, input the result to the next step.
2. Establishment and comparison of various deep learning models: four deep learning models were established and compared in this study, namely VGG19, AlexNet, CapsNet, and GoogleNet. The models using image fitting alone and those combining with clinical physical examination data were compared for each deep learning model. The diagnostic efficiency between models was expressed by the ROC curve, including AUC, F1 score, etc. the ROC curve was further analyzed by t-test, Delong test, and other statistical methods. In this study, the data were divided into a training set (70%, 30% in the training set as the validation set), and the remaining 30% as the test set to evaluate the classification accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Without any treatment before imaging examination;
2. MR of ankle joint was performed within 3 months before operation and the image quality was good;
3. Arthroscopic operation was performed in our hospital and the operation records were complete.

Exclusion Criteria:

1. history of ankle surgery, history of cancer or previous fractures.
2. Unclear image, serious artifact or incomplete clinical data.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: From September 2018 to September 2020, patients underwent ankle MRI examination in the Department of Radiology, the Third Hospital of Peking University.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Deep Learning of Anterior Talofibular Ligament: Comparison of Different Models | 2021.1-2022.3.1
  The model of deep learning was obtained for diagnosis and grading of anterior fibular ligament and compared with the doctors of different grades.

CONTACTS AND LOCATIONS:
Overall Officials: huishu Yuan, MD, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No